CLINICAL TRIAL: NCT01831076
Title: Preoperative Hormone Therapy for Postmenopausal Women With ER+ Clinical Stage T2-4 Tumors. A Phase II Study to Identify Molecular Predictors for Hormone Responsiveness and/or Resistance.
Brief Title: Preoperative Hormone Therapy for Postmenopausal Women With ER+ Clinical Stage T2-4 Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-0627.cc
Record Dates: First submitted 2013-04-04; First posted 2013-04-15 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer
Keywords: Breast cancer; estrogen receptor-positive breast cancer; progesterone receptor-positive breast cancer; Postmenopausal; Exemestane; Tamoxifen
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; 4-phenylthioandrosta-4,6-diene-3,17-dione; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (exemestane, surgery) (Active Comparator): Patients receive exemestane orally daily for 4 months in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery.
  Interventions: Drug: Exemestane
- treatment (exemestane, tamoxifen, surgery) (Experimental): Patients receive exemestane plus tamoxifen orally daily for 4 months in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery.
  Interventions: Drug: Exemestane and tamoxifen

INTERVENTIONS:
Drug: Exemestane — Given PO
  Other Names: 107868-30-4,; 6-Methyleneandrosta-1,; 4-diene-3,17-dione,; 713563,; Aromasin,; FCE 24304,; FCE-24304,; PNU 155971
  Arms: Treatment (exemestane, surgery)
Drug: Exemestane and tamoxifen — exemestane 25 mg po daily and tamoxifen 20 mg po daily given concurrently for 4 months prior to surgery
  Arms: treatment (exemestane, tamoxifen, surgery)

SUMMARY:
This phase II trial studies how well exemestane before surgery works in treating postmenopausal patients with newly diagnosed estrogen receptor positive stage II-III breast cancer. Estrogen can cause the growth of breast cancer cells. Hormone therapy using exemestane may fight breast cancer by blocking the use of estrogen by the tumor cells.

DETAILED DESCRIPTION:
This study will develop preliminary data regarding the efficacy and safety of exemestane in the preoperative treatment of postmenopausal women with ER+ or PR+ tumors. This trial is also designed to develop a predictive model to correlate expression of the known isoforms of ER and progesterone receptor (PR) and the aromatase enzyme with response to estrogenic deprivation using exemestane.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer
* ER positive (+)
* Primary tumor 2-4 regional lymph nodes 0-2 (T2-4N0-2); patients may have metastatic disease, provided local-regional surgery is clinically indicated
* Clinical stage II/III
* Postmenopausal- defined as having had a previous bilateral oophorectomy or, for women with no prior hysterectomy, the absence of spontaneous menstrual cycles for more than 1 year
* Newly diagnosed
* Patients with prior non-breast malignancies are eligible if they have been disease free for >= 5 years before study entry; patients with squamous or basal cell carcinoma of the skin that has been effectively treated, carcinoma in situ of the cervix that has been treated by surgery only, or lobular carcinoma in situ (LCIS) of the ipsilateral or contralateral breast that has been treated by surgery only are eligible, even if the cancer was diagnosed within 5 years before randomization
* Serum creatinine =< 1.5 x institutional upper limit of normal (ULN)
* Hemoglobin within normal limits for institution
* Absolute granulocyte count >= 1500
* Platelet count >= 100,000
* Serum glutamic oxaloacetic transaminase (SGOT), aspartate aminotransferase (AST) or serum glutamate pyruvate transaminase (SGPT), alanine aminotransferase (ALT) =< 2.5 x ULN
* Total bilirubin < 2 x ULN for institution
* Alkaline phosphatase < 2 x the ULN

Exclusion Criteria:

* Completely resected
* Prior hormone or chemotherapy
* Unable to take oral medication
* Patients who have nonmalignant systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude their being subjected to protocol therapy

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2002-04 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2022-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Elias, M.D, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Exemestane: Patients receive exemestane orally daily for 4 months in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery.
  Exemestane: Given PO
- Exemestane Plus Tamoxifen: preoperative exemestane plus concurrent tamoxifen for 4 months, then surgery. Patients with >T2 ER+ Her2- BC.
Period: Overall Study
Arm/Group | Exemestane | Exemestane Plus Tamoxifen
Started | 31 | 5
Completed | 30 | 4
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exemestane | Exemestane Plus Tamoxifen | Total
Number analyzed (Participants) | 31 | 5 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 4 | 22
  >=65 years | 13 | 1 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 5 | 36
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 19 | 5 | 24
  More than one race | 7 | 0 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 5 | 36

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate as Measured by Clinical Exam, Standard Imaging, and Surgical Pathology Findings
Description: Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
  Evaluated using chi-square analysis.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Exemestane | Exemestane Plus Tamoxifen
Number analyzed (Participants) | 31 | 5
Participants | 23 | 0

ADVERSE EVENTS:
Time Frame: Consent to surgery (approximately four months)
Description: Adverse event collection and reporting not required by protocol. Only SAE reporting required.
Arm/Group | Exemestane | Exemestane Plus Tamoxifen
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/5
Other Adverse Events (participants affected / at risk) | 0/31 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes